CLINICAL TRIAL: NCT02358499
Title: Genetic Variation and Variability in Posaconazole Pharmacokinetics in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1490413
Record Dates: First submitted 2015-01-29; First posted 2015-02-09 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Fungal Infections
Keywords: triazoles; fungi; transplantation, hematopoietic stem cell; leukemia; pediatrics; pharmacokinetics; bone marrow failure syndrome
MeSH Terms: conditions — Mycoses; Leukemia; Bone Marrow Failure Disorders | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Posaconazole Injection (Experimental): We will give a single dose of intravenous posaconazole and collect blood samples for pharmacokinetics (PK). The study pool will be enriched by selecting participants with known sequence variations. Every effort will be made to balance age and disease state (HSCT vs. non-HSCT).
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — Posaconazole will be given as a one time intravenous (IV) dose. The dose will take ninety (90) minutes to be infused and will be based on weight at the time of the visit.
  Other Names: Noxafil

SUMMARY:
The main goal of this study is to see how the body breaks down an antifungal drug named posaconazole in children with certain cancers, blood disorders, or transplantation of bone marrow or similar blood cells. This study will also help us learn whether a child's age, genetics, or disease affect how well the body breaks down posaconazole.

DETAILED DESCRIPTION:
The purpose of this research study is to see how the body breaks down posaconazole, which has limited data in children. Posaconazole injection has been approved by the FDA for prevention or treatment of certain fungal infections in adult patients. In children, however, we don't have data on how best to give posaconazole or whether the dosing should be personalized to individual children. This study aims to determine pharmacokinetics of posaconazole aqueous solution for injection in children aged 2 through 17 years and explores differences in drug exposure by age, genetics, and disease state. Children will receive a single dose of posaconazole injection and have their blood levels of posaconazole checked. The study will also check for safety after giving the posaconazole.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 years to under 18 years
2. Weight ≥10 kg
3. Diagnosis of any of the following: any malignancy (e.g., acute myelogenous leukemia [AML], acute lymphoblastic leukemia [ALL], lymphoma, solid tumor malignancy), hemophagocytic syndrome, bone marrow failure syndrome (e.g., myelodysplastic syndrome and aplastic anemia), hematopoietic stem cell transplantation (HSCT) recipient, or primary immune deficiency with a neutrophil or T-cell defect (e.g., chronic granulomatous disease, hyper IgE syndrome, severe combined immune deficiency).

Exclusion Criteria:

1. A female subject must not be pregnant, intend to become pregnant during the study, or breastfeed
2. A subject must not be receiving any of the following medications within 24 hours before or after posaconazole infusion (or according to standard of care protocols): sirolimus, everolimus, pimozide, quinine, HMG-CoA reductase inhibitors primarily metabolized through CYP3A4 (e.g., atorvastatin, lovastatin, simvastatin), ergot alkaloids (ergotamine, dihydroergotamine), methadone, astemizole, cisapride, halofantrine, salmeterol, or vincristine. Potential enrollees will be screened for additional concomitant medications that pose serious safety concerns when given concomitantly to posaconazole. Any of these medications will be an exclusion criterion, unless the concomitant medications may be held for 24 hours before and after posaconazole infusion or according to standard of care protocols
3. A subject must not be receiving any of the following medications concomitant (within 5 half-lives prior) to posaconazole infusion or PK sampling: rifampin, rifapentine, rifabutin, phenytoin, efavirenz, fosamprenavir, or cimetidine. Potential enrollees will be screened for additional concomitant medications that may affect posaconazole metabolism. Any of these medications will be an exclusion criterion, unless the concomitant medications may be held for 5 half-lives prior to posaconazole infusion and through PK sampling
4. A subject must not have moderate or severe liver dysfunction (except in chronic cases as judged by the P.I.) at Baseline, defined as:

   * A subject must not have moderate or severe liver dysfunction at Baseline, defined as: Aspartate aminotransferase (AST) > 5 times the upper limit of normal (ULN), OR
   * Alanine aminotransferase (ALT) > 5 times the ULN, OR
   * Serum total bilirubin >2.5 times the ULN, OR
5. A subject must not have an electrocardiogram (ECG) with prolonged age, sex-adjusted QTc interval.
6. A subject must not have a history of dysrhythmia.
7. A subject must not have creatinine clearance levels (measured or calculated) below 50 mL/min/1.73 m2.
8. A subject must not have a history of Type 1 hypersensitivity or idiosyncratic reactions to azole agents.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Posaconazole Injection | Predose on Day 1 up to 96 hours postdose
  Posaconazole concentrations in the plasma will be measured after a single dose of posaconazole injection to estimate the area under the concentration-versus-time curve (AUC). Blood samples for the assessment of AUC will be collected predose on Day 1 and then at specified time points up to 96 hours postdose.
Maximum Concentration (Cmax) of Posaconazole Injection | Predose on Day 1 up to 96 hours postdose
  Blood samples for the assessment of Cmax will be collected predose on Day 1 and then at prespecified time points up 96 hours postdose.
Time of maximum concentration (Tmax) | Predose on Day 1 up to 96 hours postdose
  Blood samples for the assessment of Tmax will be collected predose on Day 1 and then at prespecified time points up to 96 hours postdose.
Terminal half-life (t1/2) | Predose on Day 1 up to 96 hours postdose
  Blood samples for the assessment of t1/2 will be collected predose on Day 1 and then at prespecified time points up to 96 hours postdose.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (AEs) | Up to Day 4
  AEs are any unfavorable and unintended signs, symptom, or disease temporally associated with the use of a study drug, whether or nor considered related to this study drug. Treatment-emergent AEs are any event not present before starting study drug treatment or any event that was present before treatment that worsened in either intensity or frequency after exposure to study drug.
Number of Participants with Treatment-Related AEs | Up to Day 4
  AEs are any unfavorable and unintended signs, symptom, or disease temporally associated with the use of a study drug, whether or nor considered related to this study drug. Treatment-related AEs are considered by the investigator to be related to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Dwight E Yin, MD, MPH, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No